CLINICAL TRIAL: NCT00642499
Title: A Double-Blind, Randomized, Parallel-Group, Pilot Study of Oral Dronabinol Versus Placebo in the Treatment or Prevention of Highly Active Antiretroviral Therapy (HAART)-Related Nausea and Vomiting
Brief Title: Dronabinol Versus Placebo in Treatment and Prevention of Highly Active Anti-Retroviral Therapy (HAART)-Related Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Vickie Baranowski, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S175.2.101
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Highly Active Antiretroviral Therapy (HAART)-Related Nausea and Vomiting; HIV Infections
Keywords: HIV; AIDS; nausea; vomiting; HAART; Treatment Experienced; HIV Infections
MeSH Terms: conditions — Vomiting; HIV Infections; Acquired Immunodeficiency Syndrome; Nausea | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Dronabinol
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — 2.5 mg to 40 mg
  Arms: 1
Drug: Placebo — placebo
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine if dronabinol is effective in preventing or treating nausea caused by HAART (highly active anti-retroviral therapy) in HIV and AIDS patients

ELIGIBILITY:
Inclusion Criteria:

* Adherence to prior or current HAART was or is being compromised, or HAART was discontinued/interrupted due to nausea/vomiting; or beginning HAART or switching from a regimen at the time of screening for this study that did not produce significant nausea and/or vomiting to a regimen with zidovudine or a protease inhibitor (with or without low dose ritonavir).

Exclusion Criteria:

* Subjects with recent (within 30 days of randomization) or current opportunistic infection or neoplasm characteristic of AIDS (Category C of the CDC Classification System for HIV-1 infection, 1993 Revised Version).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2003-08; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The absence of nausea as indicated by a visual analog scale (VAS) score < 5 mm | 2 weeks

SECONDARY OUTCOMES:
Number of episodes vomiting/retching | 2 weeks
Duration of nausea, vomiting/retching | 2 weeks
Intensity of nausea by VAS | 2 weeks
Appetite stimulation by VAS | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (36):
- United States (36):
  - Site 911, Bakersfield, California
  - Site 919, Fresno, California
  - Site 924, Los Angeles, California
  - Site 932, Los Angeles, California
  - Site 926, Palm Springs, California
  - Site 946, Pasadena, California
  - Site 913, Tarzana, California
  - Site 907, Altamonte Springs, Florida
  - Site 948, Miami, Florida
  - Site 951, Miami, Florida
  - Site 953, Miami, Florida
  - Site 959, Miami, Florida
  - Site 954, North Palm Beach, Florida
  - Site 957, Pensacola, Florida
  - Site 923, Port Saint Lucie, Florida
  - Site 929, Sarasota, Florida
  - Site 952, Tallahassee, Florida
  - Site 931, Tampa, Florida
  - Site 908, Decatur, Georgia
  - Site 905, Boise, Idaho
  - Site 914, Chicago, Illinois
  - Site 928, Louisville, Kentucky
  - Site 955, Louisville, Kentucky
  - Site 958, New Orleans, Louisiana
  - Site 934, Boston, Massachusetts
  - Site 915, Springfield, Missouri
  - Site 956, Somers Point, New Jersey
  - Site 921, Albany, New York
  - Site 910, Cincinnati, Ohio
  - Site 941, Philadelphia, Pennsylvania
  - Site 925, Dallas, Texas
  - Site 917, Fort Worth, Texas
  - Site 906, Houston, Texas
  - Site 942, Houston, Texas
  - Site 909, Tacoma, Washington
  - Site 927, Vancouver, Washington